CLINICAL TRIAL: NCT00454324
Title: Phase II Clinical Trial of Carboplatin and Abraxane in Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Study of Abraxane and Carboplatin to Treat Small Cell Lung Cancer
Acronym: NRR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0519; CDR0000542753 (Other: PDQ number); NCT00521313 (obsolete NCT alias)
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Small Cell Lung Cancer
Keywords: Lung cancer; Small cell lung cancer; Abraxane; Paclitaxel; Carboplatin; Phase II; Randomized; Lineberger; LCCC
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Carboplatin; Albumin-Bound Paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Carboplatin + Abraxane (240mg/m2) on Day 1 of a 21 Day cycle, up to 6 cycles
  Interventions: Drug: Carboplatin; Drug: Abraxane
- Arm B (Experimental): Carboplatin + Abraxane (80mg/m2)given on Days 1, 8 and 15 of a 21 Day Cycle, up to 6 cycles
  Interventions: Drug: Carboplatin; Drug: Abraxane

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be given at a dose of target area under the concentration versus time curve in mg/mL•min (AUC)=6, on Day 1 of a 21 Day Cycle
  Other Names: Paraplatin
Drug: Abraxane — Abraxane will be given at a dose of 240mg/m2 on Day 1 of a 21 Day Cycle (Arm A)
  Abraxane will be given at a dose of 80mg/m2 on Days 1, 8, and 15 of a 21 Day Cycle (Arm B)
  Other Names: Paclitaxel

SUMMARY:
This is a phase II trial of abraxane and carboplatin in extensive stage small cell lung cancer to examine overall response rate, time to progressive disease, survival time, and assessment of toxicity profile for Carboplatin and Abraxane.

DETAILED DESCRIPTION:
Patients are being asked to be in this study because they have extensive disease small cell lung cancer. All eligible participants who agree to be in the study will receive both abraxane and carboplatin. The researchers want to evaluate the activity and safety of the combination of abraxane and carboplatin, and if this combination can help people with extensive disease small cell lung cancer.

Carboplatin is a chemotherapy drug that has been approved by the Food and Drug Administration (FDA) to treat ovarian cancer. It is in a class of drugs known as platinum-containing compounds. It slows or stops the growth of cancer cells in your body. Carboplatin is not approved by the FDA for use in the treatment of small-cell lung cancer, either alone or combined with other anti-cancer drugs. However, carboplatin given with paclitaxel is a standard or active treatment in patients with small cell lung cancer, non-small cell lung cancer, breast cancer, and ovarian cancer. Abraxane is a chemotherapy drug that was approved by the FDA to treat metastatic breast cancer after other chemotherapy has already been tried. Abraxane is a new preparation of the active ingredient in the chemotherapy drug, paclitaxel. In a study done in breast cancer patients, Abraxane was compared to paclitaxel. Abraxane has been shown to be more effective than paclitaxel in tumor response and tumor progression, in addition to having fewer side effects than paclitaxel. Abraxane was shown to cause less damage to a person's white blood cells (the cells that fight infection) and cause fewer allergic reactions; however, more patients developed numbness of their hands and feet.

Carboplatin and Abraxane are intravenous (IV) medications. Patients will begin treatment with 2 cycles (1 cycle = 21 days) of abraxane and carboplatin. Then there will be a disease assessment at cycles 2 and 4. Patients with stable disease, partial response, or complete response will get additional cycles. Patients with progressive disease no will be taken off the study treatment. A maximum of 6 cycles will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological diagnosis of extensive stage small-cell lung cancer (ES-SCLC),* including malignant pleural effusion
2. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
3. No prior systemic chemotherapy, immunotherapy, or biological therapy for SCLC
4. Measurable disease as defined by the RECIST criteria
5. Adequate organ function as defined by the protocol
6. Female patients of child bearing potential (CBP) must agree to use of reliable method of birth control during and for 3 months following treatment
7. Patients must sign informed consent document
8. Patients must be ≥ 18 years of age
9. Patients with brain metastases that have been adequately treated and are determined to be controlled by the attending physician are eligible
10. Patients who have had prior malignancies are eligible if they are ≥ 5 years from diagnosis free of disease or the attending physician believes the patient's prognosis is best defined by the ES-SCLC (if questions concerning this eligibility criteria arise, please contact the principal investigator)

(*)ES-SCLC defined as metastases outside the chest, pulmonary metastases, or contralateral metastases (supraclavicular or hilar) nodes that could not be included with a reasonable single radiation port. Patients with malignant pleural effusions are considered extensive stage.

Exclusion Criteria:

1. Received treatment within the last 30 days with a drug that has not received Food and Drug Administration (FDA) approval for any indication at the time of study entry
2. Pregnancy or breast feeding
3. Serious active infection that would require a prolonged course (4-6 weeks) of antibiotics or would compromise the safety of the patient or compromise the patient's ability to complete the study
4. Symptomatic brain metastases
5. Grade ≥ 2 neuropathy using NCI CTCAE version 3.0 criteria
6. Previous anaphylactic reaction to carboplatin, paclitaxel, and docetaxel
7. Severe or uncontrolled cardiac disease, defined as uncontrolled or unstable angina, myocardial infarction in the last month, uncontrolled congestive heart failure (≥ 3 admissions for congestive heart failure in the 3 months prior to diagnosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stinchcombe, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Grilley-Olson JE, Keedy VL, Sandler A, Moore DT, Socinski MA, Stinchcombe TE. A randomized phase II study of carboplatin with weekly or every-3-week nanoparticle albumin-bound paclitaxel (abraxane) in patients with extensive-stage small cell lung cancer. Oncologist. 2015 Feb;20(2):105-6. doi: 10.1634/theoncologist.2014-0327. Epub 2015 Jan 23. PMID 25616430
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 patients consented to participate in the study. 3 patients were consented but not treated; 2 were found ineligible, and 1 withdrew before treatment.
Groups:
- Arm A: Carboplatin + Abraxane (240mg/m2) on Day 1 of a 21 Day cycle, up to 6 cycles
  Carboplatin: Carboplatin will be given at a dose of Area Under the Curve (AUC)=6, on Day 1 of a 21 Day Cycle
  Abraxane: Abraxane will be given at a dose of 240mg/m2 on Day 1 of a 21 Day Cycle (Arm A)
  Abraxane will be given at a dose of 80mg/m2 on Days 1, 8, and 15 of a 21 Day Cycle (Arm B)
- Arm B: Carboplatin + Abraxane (80mg/m2)given on Days 1, 8 and 15 of a 21 Day Cycle, up to 6 cycles
  Carboplatin: Carboplatin will be given at a dose of AUC=6, on Day 1 of a 21 Day Cycle
  Abraxane: Abraxane will be given at a dose of 240mg/m2 on Day 1 of a 21 Day Cycle (Arm A)
  Abraxane will be given at a dose of 80mg/m2 on Days 1, 8, and 15 of a 21 Day Cycle (Arm B)
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Carboplatin + Abraxane (240mg/m2) on Day 1 of a 21 Day cycle, up to 6 cycles
  Carboplatin: Carboplatin will be given at a dose of AUC=6, on Day 1 of a 21 Day Cycle
  Abraxane: Abraxane will be given at a dose of 240mg/m2 on Day 1 of a 21 Day Cycle (Arm A)
  Abraxane will be given at a dose of 80mg/m2 on Days 1, 8, and 15 of a 21 Day Cycle (Arm B)
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Full Range); unit: years] | 70 [53 to 87] | 70.4 [60 to 80] | 70 [53 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 11 | 12
  White | 13 | 2 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Radiological imaging should be performed every 12 weeks, to ascertain the overall (or objective) response rate (Complete Response or Partial Response) according to the RECIST guidelines. Complete Response (CR) - Disappearance of all target lesions. Partial Response (PR) - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Overall Response Rate = CR+PR.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 14 | 13
percentage of participants | 79 [49 to 95] | 85 [55 to 98]

2. Secondary Outcome: 1-year Overall Survival (OS)
Description: Percentage of participants from the start of treatment with the disease that are still alive.
Time Frame: every 12 weeks for 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 14 | 13
percentage of participants | 36 [13 to 59] | 42 [15 to 67]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Defined as the time between trial enrollment to disease progression or death (whichever occurs first) or date of last contact
Time Frame: Through the end of the study, an average of approximately 8 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 14 | 13
Months | 5.8 [2.7 to 7.1] | 5.2 [2.9 to 6.7]

4. Secondary Outcome: Number of Individuals With Adverse Events
Description: Drug toxicities will be evaluated during treatment period and 30 days post treatment. Toxicities will be assessed using Common Terminology Criteria for Adverse Events (CTCAE 3.0) criteria. Grade 3 or 4 adverse events were reported
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 14 | 13
Participants
  Neutropenia | 8 | 5
  Anemia | 4 | 4
  Thrombocytopenia | 3 | 3
  Sensory neuropathy | 3 | 0
  Pain | 4 | 0
  Fatigue | 0 | 1
  Nausea | 0 | 3
  Vomiting | 0 | 2
  Diarrhea | 1 | 1

ADVERSE EVENTS:
Time Frame: Patients will be evaluated 30 days (+/- 4 days) after completion of treatment for toxicity.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 14/14 | 12/13
Serious Adverse Events (participants affected / at risk) | 7/14 | 4/13
Other Adverse Events (participants affected / at risk) | 14/14 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=14) | Arm B (N=13)
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 | 0
Pain - Esophagus (Gastrointestinal disorders) | 1 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=14) | Arm B (N=13)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 4 | 1
Alkaline phosphatase (Investigations) | 1 | 0
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 | 0
Ataxia (incoordination) (Nervous system disorders) | 1 | 0
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Creatinine (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2
Dizziness (Nervous system disorders) | 2 | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Edema: limb (General disorders) | 0 | 1
Extremity-lower (gait/walking) (General disorders) | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 | 8
Gastritis (Gastrointestinal disorders) | 0 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 | 0
Head/headache (Nervous system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 5 | 9
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Infection - Other (Specify, __) (Infections and infestations) | 1 | 0 — Infection with normal absolute neutrophil count.
Infection - Other (Specify, __) (Infections and infestations) | 0 | 1 — Right eye infection
Injection site reaction/extravasation changes (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Leukocytes (total WBC) (Investigations) | 1 | 3
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0 — Left foot drop
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 9 | 3
Neuropathy: sensory (Nervous system disorders) | 8 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 | 9
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Chest/thorax NOS (General disorders) | 1 | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Eye (Eye disorders) | 1 | 0
Pain - Head/headache (Nervous system disorders) | 1 | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Kidney (Renal and urinary disorders) | 0 | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 0 | 1
Pain - Other (Specify, __) (General disorders) | 0 | 1 — Right shoulder pain
Pain - Pain NOS (General disorders) | 1 | 0
Pain - Pelvis (Reproductive system and breast disorders) | 1 | 0
Pain - Rectum (Gastrointestinal disorders) | 0 | 1
Pain - Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pain - Stomach (Gastrointestinal disorders) | 0 | 1
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Platelets (Blood and lymphatic system disorders) | 8 | 6
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 1 | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 1
Lymphatics - Other (Specify) (Blood and lymphatic system disorders) | 1 | 0 — Lymphatics (verbatim)
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 1 | 0 — abpratpru (verbatim)
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 1 | 0
Metabolic/Lab - Other (Specify) (Metabolism and nutrition disorders) | 0 | 1 — Low total protein serum

LIMITATIONS AND CAVEATS:
The trial was closed prematurely because of slow accrual before the impact of the dose reduction on toxicity and treatment compliance could be assessed. In arm A, 6 patients required a dose reduction. In arm B, 3 patients required a dose reduction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days